CLINICAL TRIAL: NCT03478527
Title: Effects of Probiotic Bacteria on Brain Structure and Function and on Psychological Variables
Brief Title: Probiotics, Brain Structure and Psychological Variables
Acronym: ProBrain01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ProBrain01
Record Dates: First submitted 2018-01-26; First posted 2018-03-27 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Depressive Symptoms; Anxiety; Stress
Keywords: Probiotics; Psychiatric Symptoms; Cognitive Function; Hippocampus; Oxytocin; Immunological Parameters
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 1 Verum group, receiving the probiotic Vivomixx® powder
  1 Placebo group, receiving a placebo powder (similar taste and consistency as Vivomixx® powder)
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verum condition probiotics (Experimental): The verum condition probiotics in the present study is a freely available product, Vivomixx® powder (dietary supplement). Each dose (4.4g) contains 450 billion bacteria, composed of eight bacterial strains: Lactobacilli (L. paracasei, L. plantarum, L. acidophilus, L.delbrueckii subsp. bulgaricus), Bifidobacteria (B. longum, B. infantis, B. breve), and Streptococcus thermophiles. 30 Participants will be randomly assigned to this condition. The intake period is 28 days, daily dose = 4.4g.
  Interventions: Dietary Supplement: Vivomixx® powder
- placebo condition (Placebo Comparator): In the placebo condition participants will receive a placebo powder (comparable in taste and consistency to Vivomixx® = verum condition probiotics) that contains no probiotic bacteria. 30 Participants will be randomly assigned to that condition. The intake period is 28 days, daily dose = 4.4g.
  Interventions: Other: Placebo powder

INTERVENTIONS:
Dietary Supplement: Vivomixx® powder — Participants will take in a daily dose of 4.4g for 28 consecutive days
  Other Names: probiotic dietary supplement
  Arms: verum condition probiotics
Other: Placebo powder — Participants will take in a daily dose of 4.4g for 28 consecutive days
  Arms: placebo condition

SUMMARY:
Theory and research on the gut-brain-axis emphasize complex interactions between the gut microbiota, immunological and hormonal responses, brain function, brain structure, as well as resulting behavioral manifestations, such as cognitive functions and mental illness. Probiotics are living micro-organisms that change the composition of the gut microbiota and hypothetically have a positive effect on the host's general health and well-being. Probiotic bacteria naturally occur in foods such as Sauerkraut, olives, and dark chocolate, and are currently also added to industrial products such as yogurt.

Regarding the effect of probiotics on brain structure and function, animal studies have shown that the administration of probiotics in mice and rats was linked to neurogenesis in the hippocampus and an improvement of associated cognitive functions. The majority of these studies applied probiotics for 4 weeks. The substances used in these studies were often composed of several bacterial strains, suggesting that the neurogenic effect may not be reducible to a specific type of probiotic bacteria.

Probiotics seem to be effective in improving memory abilities, including spatial and non-spatial memory, both in rodents and humans. Moreover, specifically regarding the beneficial effect of probiotics on anxiety, depression and stress, preliminary evidence in humans is compelling. However methodologically sound (randomized-controlled trial [RCT], 'blind') studies are still lacking.

To sum up, the present study is going to be the first RCT with human participants that investigates structural and functional changes of the hippocampus through probiotic bacteria, using Magnet Resonance Imaging (MRI). In addition, the study aims at advancing research in the field by investigating the effects of probiotics on a broad spectrum of cognitive functions, particularly those associated with hippocampal activity (e.g. spatial memory, verbal memory). Furthermore, effects on several types of mental illness (e.g. anxiety, depression, stress) will be studied. Potential translatory mechanisms that may promote the aforementioned effects will be examined, i.e. changes in immunological parameters, 'brain derived neurotrophic factor' (BDNF), and oxytocin.

DETAILED DESCRIPTION:
A double-blind RCT intervention study will be conducted to investigate the effect of a probiotic dietary supplement vs. a placebo, taken by healthy human participants (N = 60) for 28 consecutive days. Both substances are administered in doses of 4.4g (powder) per day.

The probiotic dietary supplement used in the present study is a freely available product (in powder form) sold under the name of Vivomixx®. Per 4.4g the powder contains 450 billion bacteria, composed of eight bacterial strains: Lactobacilli (L. paracasei, L. plantarum, L. acidophilus and L.delbrueckii subsp. bulgaricus), Bifidobacteria (B. longum, B. infantis, B. breve), and Streptococcus thermophiles.

This product was chosen, because a similar supplement with an identical composition of bacteria as Vivomixx® was found to be linked to hippocampal neurogenesis in mice. The placebo powder has a similar taste and consistency as the verum (Vivomixx®) powder, but contains no probiotic bacteria.

First, participants will be screened online for eligibility (T0). Before and after the 28-day intake period, participants are asked to perform several cognitive tests and fill out questionnaires (T1, T2) at our laboratory (ca. 2 - 2.5 hours). Afterwards, blood samples will be drawn (ca. 5 minutes) and a magnet resonance tomography (MRT) session (ca. 1 - 1.5 hours) will be conducted, where participants will perform an object pattern separation task in the scanner (T1, T2). Furthermore, a follow-up after 2 months (T3), including the same assessments as at T1 and T2, will be conducted.

During the intake period participants will fill out a brief questionnaire on a weekly basis, which includes an assessment of state depression and anxiety, defecation (control item to rule out adverse effects), recent (start of) intake of medication, recent (onset of) intake of antibiotics, and recent inter-current illness (e.g. influenza). In addition, participants will record their food intake (protocol) for one week (7 consecutive days) during the intake period.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* age 18-40
* informed consent for all parts of the study (including MRT)
* none of the exclusion criteria (see below) fulfilled

Exclusion Criteria:

* age < 18 or > 40 years
* pregnancy or breastfeeding
* left-handedness
* degenerative or inflammatory diseases of the central nervous system
* severe cognitive/ neuropsychological impairment
* severe pain syndrome or other severe organic diseases
* epilepsy
* (past or present) psychiatric disorders
* neurological disorder
* severe diabetic polyneuropathy
* malignancies/ cancer
* cardiac insufficiency
* arterial hypertension
* heart attack/ stroke
* severe hepatic or renal insufficiency
* diseases of the hemopoietic system
* alcoholism/ drug addiction
* medical history of severe allergic or toxic reactions
* current participation in drug trial
* doubts about legal capacity/ capability of understanding
* referral to institutions based on court/ official order
* treatment with centrally acting medication (e.g. antipsychotics, antiepileptics, antidepressants, etc.)
* non-removable metal pieces (aneurysm clips, artificial limbs, etc.) or implanted electronic devices (pacemaker, osmotic or other implanted pumps, cochlear implants, etc.)
* claustrophobia
* acute (respiratory) infection, physical uneasiness
* tattoos in the head region, permanent make-up
* non-removable piercings
* chronic/ acute gastrointestinal diseases
* vegetarianism, veganism
* current intake of antibiotics or intake of antibiotics at any time point during the last 2 months
* lactose intolerance
* general focus on probiotic diet

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Changes in hippocampal volume, assessed via Magnet Resonance Imaging (MRI) | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in hippocampal volume in verum experimental group (in comparison to placebo control)
Changes in functional brain activation during fMRI task | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in functional connectivity (using BOLD signal) in hippocampal regions in verum experimental group (in comparison to placebo control) during pattern separation fMRI task
Changes in depression | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in levels of depression, assessed with Beck's Depression Inventory - II Revised (BDI-II-R) sum score in verum experimental group (in comparison to placebo control)
Changes in spatial navigation | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in test performance scores (number of correct responses, degree of accuracy measured as position hits) in the Tunnel task in verum experimental group (in comparison to placebo control)
Changes in Interleukin-6 (IL-6) | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in IL-6 blood serum concentration levels in verum experimental group (in comparison to placebo control)
Changes in IL-1ß | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in IL-1ß blood serum concentration levels in verum experimental group (in comparison to placebo control)
Changes in Tumor Necrosis Factor alpha (TNF-alpha) | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in TNF-alpha blood serum concentration levels in verum experimental group (in comparison to placebo control)
Changes in Brain Derived Neurotrophic Factor (BDNF) | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in blood serum level concentration of BDNF in verum experimental group (in comparison to placebo control)
Changes in verbal learning test performance | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in verbal learning performance score, assessed with the Verbal Learning Memory Test (VLMT) in verum experimental group (in comparison to placebo control)
Changes in pattern separation fMRI task | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in the pattern separation task performance (no. of correct responses to picture stimuli) in in verum experimental group (in comparison to placebo control)

OTHER OUTCOMES:
Changes in Oxytocin (OXT) | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in blood serum concentration levels of OXT in verum experimental group (in comparison to placebo control)
Changes in Processing speed or performance IQ | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in processing speed assessed by a digit-symbol test (BIS; Berliner Intelligenzskala) in verum experimental group (as compared to placebo control)
Changes in cognitive emotion regulation - functional emotion regulation | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in functional emotion regulation questionnaire sum score (as assessed with the Cognitive Emotion Regulation Questionnaire; CERQ) in verum experimental group (as compared to placebo control)
Changes in Sleepiness | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in sleepiness questionnaire sum score (ESS; Epworth Sleepiness Scale) scores in verum experimental group (as compared to placebo control)
Changes in cognitive emotion regulation - dysfunctional emotion regulation | at baseline (day 0) after intake period (day 28+) and at follow up (day 84+)
  changes in dysfunctional emotion regulation questionnaire sum score (as assessed with the Cognitive Emotion Regulation Questionnaire; CERQ) in verum experimental group (as compared to placebo control)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Kühn, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Psychiatrie und Psychotherapie, UKE Martinistraße 52, 20246 Hamburg, Germany
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buffington SA, Di Prisco GV, Auchtung TA, Ajami NJ, Petrosino JF, Costa-Mattioli M. Microbial Reconstitution Reverses Maternal Diet-Induced Social and Synaptic Deficits in Offspring. Cell. 2016 Jun 16;165(7):1762-1775. doi: 10.1016/j.cell.2016.06.001. PMID 27315483
- [Background] El Aidy S, Dinan TG, Cryan JF. Immune modulation of the brain-gut-microbe axis. Front Microbiol. 2014 Apr 7;5:146. doi: 10.3389/fmicb.2014.00146. eCollection 2014. No abstract available. PMID 24778631
- [Background] Foster JA, McVey Neufeld KA. Gut-brain axis: how the microbiome influences anxiety and depression. Trends Neurosci. 2013 May;36(5):305-12. doi: 10.1016/j.tins.2013.01.005. Epub 2013 Feb 4. PMID 23384445
- [Background] Liu J, Sun J, Wang F, Yu X, Ling Z, Li H, Zhang H, Jin J, Chen W, Pang M, Yu J, He Y, Xu J. Neuroprotective Effects of Clostridium butyricum against Vascular Dementia in Mice via Metabolic Butyrate. Biomed Res Int. 2015;2015:412946. doi: 10.1155/2015/412946. Epub 2015 Oct 7. PMID 26523278
- [Background] Liu WH, Chuang HL, Huang YT, Wu CC, Chou GT, Wang S, Tsai YC. Alteration of behavior and monoamine levels attributable to Lactobacillus plantarum PS128 in germ-free mice. Behav Brain Res. 2016 Feb 1;298(Pt B):202-9. doi: 10.1016/j.bbr.2015.10.046. Epub 2015 Oct 29. PMID 26522841
- [Background] Mohle L, Mattei D, Heimesaat MM, Bereswill S, Fischer A, Alutis M, French T, Hambardzumyan D, Matzinger P, Dunay IR, Wolf SA. Ly6C(hi) Monocytes Provide a Link between Antibiotic-Induced Changes in Gut Microbiota and Adult Hippocampal Neurogenesis. Cell Rep. 2016 May 31;15(9):1945-56. doi: 10.1016/j.celrep.2016.04.074. Epub 2016 May 19. PMID 27210745
- [Background] Wallace CJK, Milev R. The effects of probiotics on depressive symptoms in humans: a systematic review. Ann Gen Psychiatry. 2017 Feb 20;16:14. doi: 10.1186/s12991-017-0138-2. eCollection 2017. PMID 28239408
- [Background] Wang H, Lee IS, Braun C, Enck P. Effect of Probiotics on Central Nervous System Functions in Animals and Humans: A Systematic Review. J Neurogastroenterol Motil. 2016 Oct 30;22(4):589-605. doi: 10.5056/jnm16018. PMID 27413138